CLINICAL TRIAL: NCT00416819
Title: Intensive Chemotherapy and Immunotherapy in Patients With Newly Diagnosed Primary CNS Lymphoma: A Pilot Study
Brief Title: Combination Chemotherapy and Rituximab in Treating Patients With Newly Diagnosed Primary CNS Lymphoma
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000458052; UCSF-03301; UCSF-H9414-23160-02A
Record Dates: First submitted 2006-12-27; First posted 2006-12-28 (Estimated); Last update posted 2015-08-20 (Estimated); Status verified 2015-08

CONDITIONS: Brain and Central Nervous System Tumors; Lymphoma
Keywords: primary central nervous system non-Hodgkin lymphoma; primary central nervous system Hodgkin lymphoma
MeSH Terms: conditions — Central Nervous System Neoplasms; Lymphoma | interventions — Filgrastim; Rituximab; Cytarabine; etoposide phosphate; Leucovorin; Methotrexate; Temozolomide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- methotrexate, leucovorin calcium, rituximab, and temozolomide (Experimental): Determine the rate of toxicity, in terms of percentage of patients with grade 4 neurotoxicity, in patients with untreated primary CNS lymphoma treated with induction therapy comprising high-dose methotrexate, leucovorin calcium, rituximab, and temozolomide followed by consolidation therapy comprising cytarabine and etoposide phosphate.
  Interventions: Biological: filgrastim; Biological: rituximab; Drug: cytarabine; Drug: etoposide phosphate; Drug: leucovorin calcium; Drug: methotrexate; Drug: temozolomide

INTERVENTIONS:
Biological: filgrastim
Biological: rituximab
Drug: cytarabine
Drug: etoposide phosphate
Drug: leucovorin calcium
Drug: methotrexate
Drug: temozolomide

SUMMARY:
RATIONALE: Drugs used in chemotherapy work in different ways to stop the growth of cancer cells, either by killing the cells or by stopping them from dividing. Monoclonal antibodies, such as rituximab, can block cancer growth in different ways. Some block the ability of cancer cells to grow and spread. Others find cancer cells and help kill them or carry cancer-killing substances to them. Giving rituximab together with combination chemotherapy may kill more cancer cells.

PURPOSE: This clinical trial is studying the side effects and best ways to give combination chemotherapy together with rituximab in treating patients with newly diagnosed primary CNS lymphoma.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the rate of toxicity, in terms of percentage of patients with grade 4 neurotoxicity, in patients with untreated primary CNS lymphoma treated with induction therapy comprising high-dose methotrexate, leucovorin calcium, rituximab, and temozolomide followed by consolidation therapy comprising cytarabine and etoposide phosphate.

Secondary

* Determine the efficacy of this regimen, in terms of the 4-month and 12-month complete and best response rate, in these patients.
* Determine the progression-free and overall survival of patients treated with this regimen.
* Determine the percentage of patients experiencing toxicity or neurotoxicity due to this regimen.
* Determine the treatment-related mortality rate in patients treated with this regimen.
* Document the neurocognitive changes in these patients using the Mini-Mental Status Examination during the first year of treatment with this regimen.

OUTLINE: This is a pilot, multicenter study.

* Induction therapy: Patients receive high-dose methotrexate IV over 4 hours on days 1,15, 29, 43, 57, 71, and 99; leucovorin calcium IV every 6 hours on days 2-4, 16-18, 30-32, 44-46, 58-60, 72-74, and 100-102; oral temozolomide on days 7-11, 35-39, 63-67, 91-95, and 119-123; and rituximab IV on days 3, 17, 31, 45, 59, and 74. Treatment continues in the absence of disease progression or unacceptable toxicity. Patients who achieve complete response proceed to consolidation therapy.
* Consolidation therapy I: Beginning 3-4 weeks after completing induction therapy, patients receive high-dose methotrexate IV over 4 hours on day 1, leucovorin calcium IV every 6 hours on days 2-4, and oral temozolomide on days 7-11.
* Consolidation therapy II: Beginning 3-5 weeks after completing consolidation therapy I, patients receive cytarabine IV over 2 hours twice daily and etoposide phosphate IV continuously on days 1-4 and filgrastim (G-CSF) subcutaneously beginning on day 14 and continuing until blood counts recover.

After completion of study treatment, patients are followed periodically for 2 years.

PROJECTED ACCRUAL: A total of 10 patients will be accrued to this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed untreated primary CNS lymphoma (PCNSL) confirmed by 1 of the following methods:

  * Brain biopsy or resection

    * Patients diagnosed with T-cell PCNSL allowed but will not receive rituximab on study
  * Cerebrospinal fluid (CSF) cytology

    * Positive CSF cytology with or without measurable intracranial disease
  * Vitreal biopsy

    * Histologic confirmation of vitreal lymphoma with measurable intracranial tumor
* No evidence of systemic non-Hodgkin's lymphoma

  * CT scan of chest, abdomen, and pelvis or bone marrow biopsy negative for extracerebral source of lymphoma
* No evidence of pleural effusions or ascites
* MRI of brain and spine (plus gadolinium) must have measurable contrast enhancing disease unless CSF cytology is positive

PATIENT CHARACTERISTICS:

* Karnofsky performance score 50-100%
* HIV negative
* Creatinine clearance ≥ 50 mL/min
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception

PRIOR CONCURRENT THERAPY:

* No concurrent salicylates, nonsteroidal anti-inflammatory drugs, sulfonamides, or penicillins within the past week

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2003-09; Primary Completion 2005-12 (Actual); Study Completion 2012-02 (Actual)

PRIMARY OUTCOMES:
rate of toxicity in patients with untreated primary CNS lymphoma | up to 8 months
  Determine the rate of toxicity, in terms of percentage of patients with grade 4 neurotoxicity, in patients with untreated primary CNS lymphoma treated with induction therapy comprising high-dose methotrexate, leucovorin calcium, rituximab, and temozolomide followed by consolidation therapy comprising cytarabine and etoposide phosphate.

SECONDARY OUTCOMES:
Efficacy in patients with untreated primary CNS lymphoma treated with induction therapy comprising high-dose methotrexate, leucovorin calcium, rituximab, and temozolomide followed by consolidation therapy comprising cytarabine and etoposide phosphate. | up to 12 months

CONTACTS AND LOCATIONS:
Overall Officials: James L. Rubenstein, MD, PhD, Study Chair — University of California, San Francisco

REFERENCES:
- [Result] Wieduwilt MJ, Valles F, Issa S, Behler CM, Hwang J, McDermott M, Treseler P, O'Brien J, Shuman MA, Cha S, Damon LE, Rubenstein JL. Immunochemotherapy with intensive consolidation for primary CNS lymphoma: a pilot study and prognostic assessment by diffusion-weighted MRI. Clin Cancer Res. 2012 Feb 15;18(4):1146-55. doi: 10.1158/1078-0432.CCR-11-0625. Epub 2012 Jan 6. PMID 22228634